CLINICAL TRIAL: NCT01417988
Title: Prevention of Early Mortality by Presumptive TB Treatment in HIV-infected Patients Initiating Antiretroviral Therapy
Brief Title: Prevention of Early Mortality by Presumptive Tuberculosis (TB) Treatment
Acronym: PrOMPT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated prematurely due to insufficient enrolment.
Sponsor: Prof JMA Lange (Other)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor-Investigator, Prof JMA Lange, Executive Scientific Director AIGHD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIGHD_001
Record Dates: First submitted 2011-07-25; First posted 2011-08-16 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infection; Tuberculosis
Keywords: TB
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empiric TB treatment (Experimental): Empiric initiation of 4 drug TB treatment (8 weeks of 4 drug, 16 weeks of 2 drug therapy) followed by ART (efavirenz-based) within 2 weeks
  Interventions: Drug: Experimental: Empiric TB treatment
- ART only arm (Active Comparator): ART (efavirenz-based) only (+ pyridoxine 50mg) given within 2 weeks after enrolment
  Interventions: Drug: ART only arm

INTERVENTIONS:
Drug: Experimental: Empiric TB treatment — Initiation of 4 drug TB treatment (8 weeks of 4 drug, 16 weeks of 2 drug therapy) followed by ART (efavirenz-based) within 2 weeks
  Arms: Empiric TB treatment
Drug: ART only arm — ART (efavirenz-based) only (+ pyridoxine 50mg) given within 2 weeks after enrolment
  Arms: ART only arm

SUMMARY:
This study investigates the prevention of early mortality in patients initiating antiretroviral therapy (ART) in sub-Saharan Africa where 79% of the co-infected cases of TB reside. Many published studies have shown a surprisingly high proportion of all patients initiated on ART dying within 6 months (8-26%) with increasing risk with decreasing CD4 T cell count. The majority (median 70%) occur in the first 3 months with the greatest proportion of deaths due to previously undiagnosed tuberculosis (TB). The investigators will enroll patients from 4 geographically diverse countries (Gabon, Mozambique, South Africa, and Uganda) in a randomized open label clinical trial targeting a population of people with high mortality risk; patients with CD4 T cell count < 50 cells/μl and body mass index (BMI) < 18 kg/m2. Severely immunocompromised patients with low BMI in the intervention arm will receive presumptive anti-TB 4-drug chemotherapy and subsequently initiate ART within 2 weeks compared to ART alone. The main objective is to measure and compare early mortality in the group presumptively treated for TB in addition to ART. Other sub-objectives are to determine the predictors of early mortality and the causes of death by autopsy (traditional and verbal), to determine if presumptive anti-TB treatment affects viral suppression with ART, and to assess incidence rates and characterize drug toxicity in patients dually treated. Because of the high rates of TB co-infection in sub-Saharan Africa in the HIV-infected, the investigators expect that patients presumptively treated for TB in addition to HIV will have a lower mortality rate than patients receiving ART only. This trial is expected to be of great public health benefit and generalisability.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old
* HIV-1 positive
* Eligible for antiretroviral treatment with CD4 T cell count < 50 cells/μl
* BMI < 18

Exclusion Criteria:

* Patients with smear-positive pulmonary TB
* Patients who fulfill the diagnostic criteria for smear-negative pulmonary or extrapulmonary TB (http://www.who.int/tb/publications/2006/tbhiv_recommendations.pdf ).
* Previous TB treatment (history of TB medication for > 1 month
* History of using antiretroviral drugs
* Symptomatic known underlying liver disease or transaminases > 5x upper limit of normal
* Known or suspected drug resistance to more than one first-line TB drug according to WHO criteria but excluding HIV infection (e.g. household contacts of MDRTB patients)
* Pregnant or breast-feeding
* Patients with cryptococcal meningitis (CrAG positive with neurologic symptoms)
* Patients with other severe (opportunistic) disease such as disseminated KS, malignant lymphoma, toxoplasmosis who may not be able to tolerate anti-TB medication or require other specific therapy
* Patients with danger signs (respiratory rate > 30 per minute, heart rate > 120bpm, temperature > 39oC, and unable to ambulate)
* Taking other potentially life-saving medications (e.g. for other OIs, or immunosuppressants) that are incompatible with anti-TB chemotherapy or ART
* Unable to swallow TB medications
* Unable to follow-up at the clinic for regularly scheduled follow-up (e.g. too far from clinic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
All-cause mortality in the first 24 weeks after initiation of ART | 24 weeks

SECONDARY OUTCOMES:
CD4 T cell absolute increase | 24 weeks
Causes of death | 24 weeks
Safety and tolerability of anti-tuberculous medications | 24 weeks
HIV viral suppression | 24 weeks
TB incidence rates after ART initiation | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Cobelens, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Yuka Manabe, Principal Investigator — Infectious Diseases Institute at Makerere University
Locations (3):
- Medical Research Unit, Albert Schweitzer Hospital, Lambaréné, Gabon
- Ministry of Health -Provincial Heatlh Directorate of the Sofala Province (Direcção Provincial de Saúde de Sofala DPSS), Beira, Mozambique
- Infectious Diseases Institute University Makarere, Kampala, Uganda

REFERENCES:
- See also: Official Website of the sponsor — http://amc.nl